CLINICAL TRIAL: NCT00134745
Title: The Growth of Genitalia Interna and the Bone Mineralization Under Hormonal Replacement Therapy and the Presence of Aortic Root Dilatation in Girls With Turner Syndrome
Brief Title: Defining the Optimal Hormonal Replacement Therapy in Turner Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Line Cleemann (Other)
Collaborators: Novo Nordisk A/S (Industry); The County of Frederiksborg (Unknown); The foundation of Kaptajnløjtnant Harald Jensen and Wife (Unknown); The foundation of Mrs. Olga Bryde (Unknown); The foundation of Mr. Ivan Nielsen (Unknown)
Responsible Party: Sponsor-Investigator, Line Cleemann, Doctor, PhD, Hillerod Hospital, Denmark
Organization: Hillerod Hospital, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120895
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Turner Syndrome
Keywords: Turner Syndrome; Hormonal replacement therapy; Bone mineralization; Uterine size; aortic root dilatation
MeSH Terms: conditions — Turner Syndrome | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4 mg estradiol (Active Comparator)
  Interventions: Drug: estradiol
- 2 mg estradiol (Placebo Comparator)
  Interventions: Drug: estradiol

INTERVENTIONS:
Drug: estradiol — tablets, 2 mg day 1 through day 22 of the menstrual cycle for 5 years

SUMMARY:
The purpose of this study is to examine whether a larger dosage of estrogen than the one used today will secure the development of a normal sized uterus and increase the strength of the bones in girls and young women with Turner syndrome.

The purpose is also to evaluate whether aortic dilatation is present in this group of patients, and if the estrogen dosage will influence the emotional well-being and self-esteem of the patients.

DETAILED DESCRIPTION:
Turner syndrome is a common chromosomal disorder with only one X-chromosome or partial deletions in one X-chromosome in all or some of the cell-lines in the body. Appr. 18 girls/year are being born with the syndrome in Denmark. The syndrome is mostly known for reduced final height and the lack of pubertal development with infertility, but it is also known for diseases influencing other parts of the body like the heart with the risk of development of aortic dilatation and subsequently dissection with the risk of rupture, profuse bleeding and sudden death. Reduced bone strength and increased risk of bone fracture are also features of the syndrome. Treatment with growth hormone and female sex-hormones are well-established treatments.

Girls and young women with Turner syndrome ages 10 to 21 years will participate. The girls ages 15 to 21 years will randomly and double blindly receive treatment with either 2 mg or 4 mg estrogen for 5 years. Yearly examinations with blood tests, physical examinations, questionnaires, ultrasound and MR-scan of the internal female genitalia, DEXA-scan of the bones and MR-scan of the heart will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Verified Turner syndrome
* Ages 10-25 years

Exclusion Criteria:

* Contraindications to the MR-scan
* Contraindications to the trial medication
* Severe or chronic sickness with impact on the parameters of the study or incompatibility with the trial medication
* Intake of medications with interactions with trial medication

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2005-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The size of the uterus evaluated by magnetic resonance (MR)-scan | 5 years
Bones evaluated by dual-energy X-ray absorptiometry (DEXA)-scan | 5 years

SECONDARY OUTCOMES:
The diameter of the aortic root evaluated by MR-scan | 5 years
Development of biochemical markers | 5 years
Body composition evaluated by DEXA-scan | 5 years
Emotional wellbeing and self-esteem evaluated by questionnaires | 5 years
The size of the uterus evaluated by ultrasound | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Line Cleemann, Doctor, Principal Investigator — Pediatric Unit, Hillerod Hospital
Locations (1):
- Pediatric Unit, Hillerod Hospital, Hillerød, Frederiksborg County, Denmark

REFERENCES:
- [Derived] Cleemann L, Holm K, Fallentin E, Moller N, Kristensen B, Skouby SO, Leth-Esbensen P, Jeppesen EM, Jensen AK, Gravholt CH. Effect of Dosage of 17ss-Estradiol on Uterine Growth in Turner Syndrome-A Randomized Controlled Clinical Pilot Trial. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz061. doi: 10.1210/clinem/dgz061. PMID 31613320
- [Derived] Brun S, Cleemann L, Holm K, Salskov G, Erlandsen M, Berglund A, Andersen NH, Gravholt CH. Five-Year Randomized Study Demonstrates Blood Pressure Increases in Young Women With Turner Syndrome Regardless of Estradiol Dose. Hypertension. 2019 Jan;73(1):242-248. doi: 10.1161/HYPERTENSIONAHA.118.11742. PMID 30571546